CLINICAL TRIAL: NCT01255475
Title: Effect of Blood Pressure Reduction in Patients With Chronic Heart Failure - Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Blood Pressure Reduction in Heart Failure
Acronym: REPIC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Edimar Alcides Bocchi, Heart Failure Team Directos, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNPq 474992/2009-8
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure; Cardiac Failure; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Hydralazine; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: Hydralazine/amlodipine
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydralazine/amlodipine — Patients will receive drug therapy aimed to reducing blood pressure - first line drug will be hydralazine up to 100mg/day; if systolic blood pressure reduces less than 20% from baseline and remains over 100mmHg patients will further receive amlodipine up to 10mg/day
  Arms: Intervention
Drug: Placebo — Patients will receive placebo
  Arms: Control

SUMMARY:
Previous studies have demonstrated a direct association between blood pressure level and cardiovascular risk. However in patients with heart failure this association is considered controversial. The aim of this study is to evaluate the effect of the reduction of blood pressure in patients with heart failure. The investigators will examine the effects of this intervention over mortality, quality of life, and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic heart failure for at least 6 months
* ejection fraction of 40% or less, as measured by transthoracic echocardiography
* optimal clinical treatment for chronic heart failure according to current international guidelines.

Exclusion Criteria:

* patient refusal
* rheumatic or degenerative valvular disease
* restrictive cardiomyopathy
* evidence of myocardial ischemia
* alcohol or drug use
* malignant neoplasm
* active infection
* surgical intervention in the 3 previous months
* lactation, childbearing or childbearing potential.
* pulmonary embolism in the 6 previous months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Any cause mortality | 12 months after randomization
Unplanned hospital admission from any cause | 12 months after randomization

SECONDARY OUTCOMES:
Cardiovascular death | 12 months after randomization
Acute myocardial ischemia | 12 months after randomization
Stroke | 12 months after randomization
Symptomatic hypotension | 12 months after randomization
Renal function | 12 months after randomization
Peak exercise oxygen consumption | 12 months after randomization
Quality of life | 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Edimar A Bocchi, Prof., Principal Investigator — Heart Institute (InCor) HC FMUSP
Locations (1):
- Heart Institute (InCor) do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil